CLINICAL TRIAL: NCT05086523
Title: Addendum to Protocol CS-03: Clinical Evaluation of Safety and Effectiveness of the BackBeat Medical Moderato System in Patients With Hypertension: A Double-Blind Randomized Trial, NCT02837445
Brief Title: Cardiac Neuromodulation Therapy (CNT) "Washout" Sub-Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BackBeat Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CNT Washout substudy
Record Dates: First submitted 2021-09-27; First posted 2021-10-21 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Hypertension,Essential; Systolic Hypertension
MeSH Terms: conditions — Essential Hypertension; Isolated Systolic Hypertension

STUDY DESIGN:
Intervention Model Description: each patient serves as his/her own control, in the PHC ON (baseline) to OFF transition (early time point), then a week later again, the OFF value (late time point) will be compared to baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Programmable Hypertension Control (BackBeat Moderato) — Programmable Hypertension Control can be turned OFF without affecting regular pacing
Device: Pacing (BackBeat Moderato) — Programmable Hypertension Control can be turned OFF without affecting regular pacing

SUMMARY:
This washout protocol is structured as a sub-study for patients willing to participate after finishing the double blind randomised phase of the clinical trial, NCT02837445. Devices will be turned off for a week approximately. Patients will have their PHC programmed to automatically turn off 24 hr after a medical and technical visit and remain in regular pacing. Ambulatory recording of the BP will start at the end of the visit, and continue for 24 hr after the turn off time (48 hr recording). Conversely, patients will return at the end of the first week, when a second 48 hr recording will be initiated, this time, the PHC will be programmed to turn on 24 hr later. The recordings therefore will provide data of the ON to OFF transition for the evaluation of the residual effect of PHC after 24 h and after week.

DETAILED DESCRIPTION:
As detailed in protocol CS-03, the BackBeat Moderato system applies standard pacing signals according to a specially timed, alternating sequence short and longer atrioventricular (AV) delays, to reduce blood pressure as a treatment for hypertension. The algorithm that governs the delivery of these pacing signals is referred to as Cardiac Neuromodulation Therapy (CNT) and the signals are referred to as Programable Hypertension Control (PHC) signals, (refer to Clinical Evaluation of Safety and Effectiveness of the BackBeat Medical Moderato System in Patients With Hypertension: A Double-Blind Randomized Trial, NCT02837445) As currently used, CNT requires continuous right ventricle (RV) pacing. However, due to potentially long-term effects of CNT on baroceptor function, intermittent deactivation of CNT could reduce the overall amount of pacing without loss of efficacy. Support for this hypothesis comes from a preclinical testing of CNT that was detailed in "Chapter II - Pre-Clinical Testing" of the approved Investigator Brochure. BackBeat Medical conducted a chronic feasibility study in 4 dogs with hypertension induced by renal artery banding which were implanted with a Moderato IPG for 4 months. Results from this study showed that when CNT was turned off after 30 days of continuous CNT, there was a very slow increase in systolic pressure, approaching pre-therapy levels only several weeks later. A 50% residual effect remained at 20 days, with a total washout period of approximately 30 days.

One possible explanation for this observation is that the signal beneficially changes the pressure"set point" of the baroceptor reflexes. Changes in the set point could result from changes at the level of either the pressure sensor in the carotid sinus or within the pressure regulatory region of the central nervous system; namely the nucleus tractus solitarius (NTS) in the medulla oblongata.

This sub-study aims to evaluate whether and for how long the blood-pressure lowering effect of CNT persists following its cessation in patients who have been treated with CNT for a prolonged period of time.

ELIGIBILITY:
Inclusion Criteria:

* Subject is implanted with a Moderato® implantable pulse generator (IPG) and is being followed by the site per standard of care.
* Subject has an average office systolic blood pressure > 130 mmHg and < 170 mmHg at the sub-study screening visit.

Exclusion Criteria:

* Subject has permanent atrial fibrillation.
* Subject had significant paroxysmal atrial fibrillation/flutter burden (defined as >25% of beats) in the past month. Atrial fibrillation/flutter burden will be determined by interrogation of the Moderato pulse generator.
* Subject experienced neurological events (stroke or TIA) within the past year. Subject have had a serious adverse event classified as related to CNT or the Backbeat Moderato device.
* Female subject who is pregnant, breast-feeding, intends to become pregnant or has the possibility of becoming pregnant during the conduct of the study and is not willing to use contraception during the study.
* Subject cannot or is unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) between baseline (PHC ON) and PHC OFF at two consecutive time points: (a) after one day and (b) after a week of PHC OFF | one week
  The first 24 hr of the first recording will be used to obtain the average for the baseline SBP value. As PHC is automatically turned OFF while the recording continues for another 24 hrs, the latter 24 hr will be used to obtain the average SBP of the first day with PHC OFF. A week later, the first 24 hr of the second recording will be used to obtain the average change in SBP to compare to the baseline (PHC ON).

CONTACTS AND LOCATIONS:
Locations (6):
- Na Homolce Hospital, Prague, Czechia
- Semmelweis University Heart and Vascular Center, Budapest, Hungary
- Poland (4):
  - Szpital Kliniczny Przemiemienia Panskiego, Poznan
  - Pomeranian Medical University Hospital no. 2, Szczecin
  - Samodzielnym Publicznym Centralnym Szpitalem Klinicznym, Warsaw
  - Silesian Center for Heart Diseases, Zabrze

REFERENCES:
- [Background] Kandzari DE, Kario K, Mahfoud F, Cohen SA, Pilcher G, Pocock S, Townsend R, Weber MA, Bohm M. The SPYRAL HTN Global Clinical Trial Program: Rationale and design for studies of renal denervation in the absence (SPYRAL HTN OFF-MED) and presence (SPYRAL HTN ON-MED) of antihypertensive medications. Am Heart J. 2016 Jan;171(1):82-91. doi: 10.1016/j.ahj.2015.08.021. Epub 2015 Sep 11. PMID 26699604
- [Background] Bohm M, Townsend RR, Kario K, Kandzari D, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Hickey GL, Fahy M, DeBruin V, Brar S, Pocock S. Rationale and design of two randomized sham-controlled trials of catheter-based renal denervation in subjects with uncontrolled hypertension in the absence (SPYRAL HTN-OFF MED Pivotal) and presence (SPYRAL HTN-ON MED Expansion) of antihypertensive medications: a novel approach using Bayesian design. Clin Res Cardiol. 2020 Mar;109(3):289-302. doi: 10.1007/s00392-020-01595-z. Epub 2020 Feb 7. PMID 32034481
- [Background] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944